CLINICAL TRIAL: NCT05523167
Title: A Phase 2/3, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Group, 2-Arm, Multicenter, Operationally Seamless Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Efgartigimod PH20 SC in Participants Aged 18 Years and Older With Active Idiopathic Inflammatory Myopathy
Brief Title: A Study to Investigate the Efficacy and Safety of Efgartigimod PH20 SC in Adult Participants With Active Idiopathic Inflammatory Myopathy.
Acronym: ALKIVIA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARGX-113-2007; 2024-512785-33-00 (EU CTIS Number)
Record Dates: First submitted 2022-08-30; First posted 2022-08-31 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Active Idiopathic Inflammatory Myopathy; Myositis; Dermatomyositis; Polymyositis; Immune-Mediated Necrotizing Myopathy; Antisynthetase Syndrome
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Antisynthetase syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EFG PH20 SC (Experimental): participants receiving efgartigimod PH20 SC on top of background treatment
  Interventions: Biological: EFG PH20 SC
- PBO PH20 SC (Placebo Comparator): participants receiving placebo PH20 SC on top of background treatment
  Interventions: Other: PBO

INTERVENTIONS:
Biological: EFG PH20 SC — Subcutaneous injection of efgartigimod coformulated with rHuPH20, a permeation enhancer
  Arms: EFG PH20 SC
Other: PBO — Subcutaneous injection of placebo coformulated with rHuPH20, a permeation enhancer
  Arms: PBO PH20 SC

SUMMARY:
This study's purpose is to measure the treatment response from efgartigimod PH20 SC compared with placebo in participants with Idiopathic Inflammatory Myopathy (IIM). Participants with the IIM subtypes of dermatomyositis (DM), immune-mediated necrotizing myopathy (IMNM), or certain other subtypes of polymyositis (PM; including antisynthetase syndrome [ASyS]) will be included in the study. Treatment response will be measured by Total improvement score (TIS). Additional information can be found on https://myositis-study.com/.

ELIGIBILITY:
Inclusion Criteria:

* Ability to consent in the jurisdiction in which the study is taking place and capable of giving signed informed consent.
* A definite or probable clinical diagnosis of idiopathic inflammatory myopathy (IIM)
* One of the following medical histories: Diagnosis of dermatomyositis (DM) or juvenile dermatomyositis (JDM), Diagnosis of polymyositis (PM) (including antisynthetase syndrome (ASyS)), Diagnosis of immune-mediated necrotizing myopathy (IMNM)
* Diagnosed with active disease as defined by the presence of at least 1 of the following criteria: Abnormal levels of at least 1 of the following enzymes: creatine kinase (CK), aldolase, lactate dehydrogenase, aspartate aminotransaminase (AST), alanine aminotransferase (ALT), based on central laboratory results; Electromyography demonstrating active disease within the past 3 months; Active dermatomyositis (DM) skin rash; Muscle biopsy indicative of active idiopathic inflammatory myopathy (IIM) in the past 3 months; Magnetic resonance imaging within the past 3 months indicative of active inflammation
* Muscle weakness
* Receiving a permitted background treatment for idiopathic inflammatory myopathy.
* Contraceptive use consistent with local regulations, where available, for individuals participating in clinical studies. Women of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test at baseline before receiving investigational medicinal product (IMP).

The full list of inclusion criteria can be found in the protocol.

Exclusion Criteria:

* A clinically significant active infection at screening
* A COVID-19 polymerase chain reaction (PCR)-positive test before enrollment
* Any other known autoimmune disease that, in the investigator's opinion, would interfere with an accurate assessment of clinical symptoms of idiopathic inflammatory myopathy (IIM) or put the patient at undue risk
* A history of malignancy unless considered cured by adequate treatment, with no evidence of recurrence for ≥ 3 years before the first administration of the investigational medicinal product (IMP). Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer ; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological finding of prostate cancer
* Severe muscle damage
* Glucocorticoid-induced myopathy that the investigator considers the primary cause of muscle weakness or permanent weakness linked to a non-idiopathic inflammatory myopathy (IIM) cause
* Juvenile myositis (JDM) diagnosed > 5 years from screening or juvenile myositis with extensive calcinosis or severe calcinosis.
* Uncontrolled interstitial lung disease or any other uncontrolled idiopathic inflammatory myopathy (IIM) manifestation that, in the opinion of the investigator, would be likely to require treatment with prohibited medication during the study
* Other inflammatory and noninflammatory myopathies: inclusion body myositis, overlap myositis), metabolic myopathies, muscle dystrophies or a family history of muscle dystrophy, drug-induced or endocrine induced myositis, and juvenile myositis (other than juvenile dermatomyositis (JDM))
* Clinically significant disease, recent major surgery or intends to have surgery during the study, or has any other condition in the opinion of the investigator that could confound the results of the trial or put the patient at undue risk
* Known hypersensitivity reaction to investigational medicinal product (IMP) or 1 of its excipients
* Received a live or live-attenuated vaccine less than 4 weeks before screening.
* Positive serum test at screening for active viral infection with any of the following conditions: Hepatitis B virus (HBV); Hepatitis C virus (HCV); HIV
* Participant has previously participated in an efgartigimod clinical trial and received at least 1 dose of investigational medicinal product (IMP).
* Participant is concurrently participating in any other clinical study, including a noninterventional study.
* Participant has a current or history (ie, within 12 months of screening) of alcohol, drug, or medication abuse.
* Participant is pregnant or lactating or intends to become pregnant during the study.
* Participant has severe renal impairment .
* Participant is institutionalized by a court or other governmental order or is in a dependent relationship with the sponsor or investigator.

The full list of exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Total improvement score (TIS); measured on a [0,100] scale. Higher scores represent improvement; zero indicates no improvement or worsening (from baseline). | phase 2: 24 weeks; phase 3: 52 weeks

SECONDARY OUTCOMES:
Time to reach TIS ≥ 20 (first "minimal clinical improvement") | phase 2: up to 24 weeks; phase 3: up to 52 weeks
Percentage of participants with TIS ≥ 20 | phase 2: 24 weeks; phase 3: 52 weeks
Time to reach TIS ≥ 40 (first "moderate clinical improvement") | phase 2: up to 24 weeks; phase 3: up to 52 weeks
Percentage of participants with TIS ≥ 40 | phase 2: 24 weeks; phase 3: 52 weeks
Change in manual muscle testing-8 (MMT8) score | phase 2: 24 weeks; phase 3: 52 weeks
Change in Patient Global Assessment of Disease Activity (PGA) | phase 2: 24 weeks; phase 3: 52 weeks
Change in Physician Global Assessment of Disease Activity (MDGA) | phase 2: 24 weeks; phase 3: 52 weeks
Proportion of participants achieving target dose of ≤ 5 mg (prednisone equivalent) | Phase 3: 52 weeks

CONTACTS AND LOCATIONS:
Locations (202):
- United States (40):
  - Neuromuscular Research Center, Phoenix, Arizona
  - HonorHealth Neurology - Bob Bove Neuroscience Institute - Neurology, Scottsdale, Arizona
  - Attune Health Research, Inc, Beverly Hills, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Profound Research LLC - Oceanside, Oceanside, California
  - University of California, Irvine, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Stanford Medicine Outpatient Center - Stanford Dermatology Clinic-Stanford University School of Medicine, Redwood City, California
  - California Pacific Medical Center - Sutter Health, San Francisco, California
  - Amyotrophic Lateral Sclerosis (ALS) Treatment Center,University of California San Francisco (UCSF), San Francisco, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Yale Cancer Center-Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - UF Health Rheumatology, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida (USF) - Morsani Center (USF Health Carol and Frank Morsani Center for Advanced Healthcare), Tampa, Florida
  - Emory University Hospital, The Emory Clinic, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Medicine - Johns Hopkins Myositis Center, Baltimore, Maryland
  - Harvard Medical School - Brigham and Women's Hospital (BWH) - The Schuster Family Transplantation Research Center (TRC), Boston, Massachusetts
  - Michigan State University - Neurology, East Lansing, Michigan
  - St. Paul Rheumatology, PA, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Great Neck, New York
  - Hospital for Special Surgery, New York, New York
  - University of North Carolina (UNC) School of Medicine, Chapel Hill, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Mercy Hospital - Mercy Clinic Neurology Oklahoma City - Neurology, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center (VUMC) - Vanderbilt Rheumatology Clinic, Nashville, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - McGovern Medical School -The University of Texas Health Science Center at Houston, Houston, Texas
  - Nerve And Muscle Center Of Texas, Houston, Texas
  - University of Vermont Medical Center - Main Campus, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
- Argentina (5):
  - Consultora Integral de Salud, Córdoba
  - Framingham Centro Medico, La Plata
  - Dim Clinica Privada, Ramos Mejía
  - Centro Dermatologico Schejtman, San Miguel
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Australia (2):
  - The Wesley Medical Research, Auchenflower
  - Fiona Stanley Hospital, Murdoch
- Austria (2):
  - Medical University Innsbruck, Innsbruck
  - Allgemeines Krankenhaus der Stadt Wien (AKH Wien), Vienna
- Belgium (4):
  - Centre Hospitalier Universitaire de Charleroi, Charleroi
  - AZ Sint Lucas Gent-Campus Sint Lucas, Ghent
  - Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- Bulgaria (2):
  - Medical Centre Artmed, Plovdiv
  - Multiprofile hospital for active treatment Kaspela EOOD, Plovdiv
- Canada (2):
  - Genge Partners, Montreal
  - Ottawa Hospital Research Institute-Civic Campus, Ottawa
- China (20):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital - School of Medicine - ZheJiang University, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital Of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Renji Hospital, Shanghai
  - First Affiliated Hospital of Shanxi Medical College, Shanxi
  - China Medical University (CMU) - First Affiliated Hospital, Shenyang
  - Huazhong University of Science and Technology - Tongji Medical College - Tongji Hospital, Wuhan
  - First Affiliated Hospital (Henan Medical University - First Affiliated Hospital)-Zhengzhou University, Zhengzhou
- Cyprus Institute of Neurology and Genetics, Nicosia, Cyprus
- Revmatologicky ustav, Prague, Czechia
- Copenhagen University Hospital-Rigshospitalet University Hospital, Copenhagen, Denmark
- France (4):
  - Hopital Edouard Herriot, Lyon
  - Reference Center Neuro-Muscular Diseases - CHU Paris Group Hospitalier La Pitie Salpetriere-Charles Foix, Paris
  - Centre Hospitalier Universitaire (CHU) Hopitaux de Rouen, Rouen
  - Hopitaux Universitaire de Strasbourg-Centre de References des Maladies Autoimmunes, Strasbourg
- Georgia (6):
  - American Hospital Network, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Aversi Clinic, Tbilisi
  - LLC MediClub Georgia, Tbilisi
  - The First Medical Center, Tbilisi
  - LTD Tbilisi Heart Center, Tbilisi
- Germany (10):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitatsmedizin Gottingen - Georg-August-Universitat, Göttingen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitatsmedizin Mannheim, Mannheim
  - Ludwig-Maximilians-Universitat Munchen Friedrich-Baur-Institut Neurologische Klinik und Poliklinik, München
  - St. Josef-Stift Sendenhorst, Sendenhorst
  - Universitaetsklinikum Tuebingen (UKT), Tübingen
  - Universitatsklinikum Ulm - Standort Oberer Eselsberg, Ulm
- Greece (5):
  - National and Kapodistrian University of Athens - School of Health Sciences - Faculty of Medicine, Athens
  - National and Kapodistrian University of Athens - Eginition Hospital, Athens
  - Attikon General University Hospital, Athens
  - Athens Medical Center, Athens
  - University of Ioannina Medical School, Ioannina
- Hungary (2):
  - Semmelweis Egyetem, Institute of Genomic Medicine and Rare Disorders, Budapest
  - Debreceni Egyetem - University of Debrecen, Debrecen
- Ireland (3):
  - St. Vincents University Hospital, Dublin
  - Connolly Hospital Blanchardstown, Dublin
  - North West Rheumatology Unit - Our Lady's Hospital, Manorhamilton
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Beilinson Campus (Beilinson and Hasharon Hospital), Petah Tikva
  - Sheba Medical Center - Rheumatology, Ramat Gan
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Consorziale Di Bari - Rheumatology, Bari
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele Hospital, Milan
  - San Matteo Hospital, Pavia
  - A.O. Universitaria Pisana, Pisa
  - IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - IRCCS Istituto Clinico Humanitas - Rheumatology, Rozzano
  - Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino - Presidio Molinette, Torino
  - ASU FC - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Japan (18):
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyō City
  - Nippon Medical School - Nippon Medical School Hospital, Bunkyō City
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Kurume University Hospital, Kurume
  - Chiba-Nishi General Hospital, Matsudo-shi
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya
  - Kitasato University Hospital (KUH), Sagamihara-shi
  - Sapporo City Hospital, Sapporo
  - Hokkaido University Hospital - Rheumatology, Sapporo
  - Sasebo Chuo Hospital, Sasebo-shi
  - Tohoku University Hospital, Sendai
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital - Rheumatology, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - University of Tsukuba Hospital - Rheumatology, Tsukuba
  - Yamaguchi University Hospital, Ube-shi
  - Wakayama Medical University Hospital - Dermatology, Wakayama
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (2):
  - CITER - Centro de Investigacion y Tratamiento de las Enfermedades Reumaticas S.A. de C.V., Mexico City
  - Centro Peninsular De Investigacion Clinica, Mérida
- Netherlands (2):
  - Amsterdam University Medical Center (Amsterdam UMC), Academic Medical Center (AMC), Amsterdam
  - Universitair Medisch Centrum Utrecht (UMC Utrecht), Utrecht
- Peru (4):
  - Hogar Clinica San Juan de Dios, Arequipa
  - Investigaciones Clinicas S.A.C., Lima
  - Instituto Peruano Del Hueso Y La Articulacion Sac-Privado-Lima, Centro De Investigacion Iphar, Lima
  - Hospital Nacional Cayetano Heredia, Lima
- Poland (3):
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - USK-WAM Centralny Szpital Weteranow - Szpital Kniniczny ul. Zeromskiego 113, Lodz
  - Centrum Wsparcia Badan Klinicznych Pomorski Uniwersytet Medyczny w Szczecinie, Szczecin
- Portugal (2):
  - Centro Hospitalar Lisboa Norte, E.P.E- Hospital Santa Maria, Lisbon
  - Centro Hospitalar Universitario de Santo Antonio, Porto
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Institute of Rheumatology, Belgrade
- Narodny ustav reumatickych chorob, Piešťany, Slovakia
- South Korea (6):
  - Chungnam National University Hospital (CNUH), Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (9):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona - Sede Villarroel - Rheumatology, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital De Valme, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Do Meixoeiro, Vigo
- Karolinska Universitestssjukhus Solna, Stockholm, Sweden
- Neurocenter of Southern Switzerland, Lugano, Switzerland
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University and Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
- Thailand (7):
  - Chulalongkorn University - Faculty of Medicine - King Chulalongkorn Memorial Hospital (KCMH), Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi hospital, Bangkok
  - Siriraj Hospital, Mahidol University of Internal medicine, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty, Ankara
  - Ankara City Hospital, Ankara
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- United Kingdom (9):
  - Royal National Hospital for Rheumatic Diseases - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Doncaster Royal Infirmary - Doncaster And Bassetlaw Hospitals Nhs Foundation Trust, Doncaster
  - Leeds Institute of Rheumatic & Musculoskeletal Medicine - University of Leeds, Leeds
  - Aintree University Hospital - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - The Royal Free Hospital - Royal Free London NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - The National Hospital for Neurology and Neurosurgery, London
  - James Cook University Hospital - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Salford Royal Hospital, Northern Care Alliance NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://myositis-study.com/